CLINICAL TRIAL: NCT00208585
Title: A Randomized Placebo-Controlled Trial of Sertraline for the Neurobehavioral Sequelae of Traumatic Brain Injury
Brief Title: Sertraline vs. Placebo for Symptoms Following Traumatic Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: The Defense and Veterans Brain Injury Center (U.S. Federal Agency); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); VA Palo Alto Health Care System (U.S. Federal Agency); Hunter Holmes McGuire VA Medical Center (U.S. Federal Agency); United States Naval Medical Center, San Diego (U.S. Federal Agency); James A. Haley Veterans Administration Hospital (U.S. Federal Agency); 59th Medical Wing (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00-7102
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Sertraline

INTERVENTIONS:
Drug: sertraline

SUMMARY:
The purpose of this study is to investigate the efficacy of an SSRI, sertraline for the use of post-concussive symptoms following a traumatic brain injury. the study also seeks to investigate the relationship between irritability and aggression and anosmia in individuals who have suffered a traumatic brian injury.

DETAILED DESCRIPTION:
The objectives of this protocol are the following:

1. To investigate the efficacy of sertraline, a selective serotonin reuptake inhibitor (SSRI), in treating neurobehavioral sequelae of irritability, depression, frustration, anxiety and other post-concussive symptoms following traumatic brain injury (TBI).
2. To explore possible relationships between anosmia (deficits in smell) and irritability/ aggression.

This study will test the hypotheses:

Sertraline is effective in treating Post TBI neurobehavioral symptoms of irritability, depression, frustration, anxiety, and other elements of the postconcussive syndrome.

Patients who receive sertraline will have significantly less post-concussive symptoms at 12 weeks than patients who received placebo. Post-concussive symptoms will be measured by the Gouvier Post-Concussive Syndrome Scale (PCSC) and the Affective Cluster score of the Cicerone Post Concussive Scale.

Patients with anosmia will have greater irritability and aggressive symptoms than those without anosmia.

. Subjects: One hundred people will take part in this study: approximately 50 subjects will take sertraline and 50 will take placebo. These patients will be selected from referrals to the Defense and Veterans Head Injury Program at WRAMC. Patients will be active duty or other military beneficiaries, between 18 and 65 years of age. Males and non-pregnant females may participate.

b. Inclusion and Exclusion Criteria:

1. Inclusion:

   1. Traumatic brain injury patients within 6 months of injury.
   2. Traumatic brain injury with:

      Minimum severity - TBI with post traumatic amnesia. Maximum severity - recovery to a Rancho los Amigos (see Appendix II) level 7 or 8 by six months after injury.
   3. The C Criterion of DSM IV diagnosis of Post Concussive Disorder (PCD- Research Criteria), with symptoms persisting for a minimum of 4 weeks.
   4. Military beneficiary.
2. Exclusion criteria:

   1. Severe prior neurologic or psychiatric illness, such as stroke or psychosis. (Previous nonpsychotic depression is not an exclusion criterion)
   2. Contraindication to the use of sertraline.
   3. Previous severe traumatic brain injury (defined as TBI with period of unconsciousness greater than 1 week prior. This exclusion refers only to TBI's prior to the current injury, which is within the past 6 months).
   4. Pregnancy
   5. Current active suicidal ideation

   c. Study Design: This study will be a prospective, double-blind, randomized 1:1 control trial study with two groups: active drug and placebo. Block randomization will be used so neither the patient nor the study physician will be able to guess the study drug assignment.

   d. Methodology: Patients will receive a multidisciplinary evaluation consisting of neurology exam, neuropsychology, psychiatry, speech and language, psychosocial, rehabilitation medicine (FIM/FAM), EEG, MRI, phlebotomy, and family interview. Blood samples will be kept at the DVHIP labeled with the patient's study number for possible future use in studies to better understand recovery from head injury. No studies would be performed on the blood samples until the patients have signed an additional informed consent with additional details on the blood studies planned. After signing the volunteer informed consent for the current sertraline protocol, evoked potentials and the smell test ( see Appendix III) will be administered and patients will be randomized into an active drug or placebo group. Patients will receive an increasing dose of sertraline or placebo up to a dose of 200 mg of sertraline. See Table I, Appendix I, for dosing schedule. All patients will receive a two part counseling session regarding brain injury and recovery from brain injury. The first session will cover the types of symptoms that may be experienced after brain injury, the expected course of recovery, and recommendations for symptom management. The second will begin with a brief assessment of material retained from the first counseling session, and continue with specific recommendations that match general principles to the patient's specific life situation. A brief pre-test and post-test (see Appendix IV) on general TBI information will be given with the first counseling session; a pre-test will be administered prior to the second session. These tests will permit better understanding of how much information patients have regarding TBI and how much is retained after a first counseling session.

   The medication phase will last 12 weeks. Patients will receive standard TBI care during this period. Current standard of care for patients with moderate-severe TBI following a full evaluation with medical/surgical treatment of any acute medical/surgical conditions is approximately 8 weeks of Convalescent Leave Home (CVL) followed by a gradual return to duty. Mild TBI patients typically receive 1-4 weeks of CVL followed by a gradual return to duty. Civilians would have similar schedules for resumption of activities. From current referral patterns, we expect most patients to have moderate traumatic brain injuries. The DVHIP experience suggests that patients are virtually never referred to DVHIP severely depressed and already on therapeutic levels of antidepressants. More commonly, patients are referred with mild-moderate symptoms of sleep difficulties, headache, irritability and/or depression. Because no randomized, controlled trials exist to suggest that current medical treatment is effective in these patients, and because a substantial placebo effect is a known reality, the design of this study (randomization to sertraline or placebo) is appropriate. Also, we have cared for a few patients who, although clinically depressed, refused medications. We worked with them in a supportive educational framework, and in some cases, their depressions remitted. Thus, the best treatment for these patients is far from established. It is likely that future research will help clarify which treatments are best for which patients. For this study, patients who may have been started on a tricyclic antidepressant (e.g., for headache) or an SSRI will be withdrawn from these medications for 10 days prior to the start of the study medication. Patients will be informed of concomitant medication options if the test article (sertraline or placebo) is not sufficient for treating their symptoms, or if they feel they need medication prior to the start of the test article. All patients will be contacted weekly during the medication phase to assess general condition, current symptoms, and assessment of compliance. Patients will be rated for improvement at weeks 3, 6, and 9 for possible medication adjustment. The determination of medication adjustment will be made by study personnel at Walter Reed only. If patients require a clinical medical appointment during the 12 weeks, patients will be seen at WRAMC if possible. If not possible, study personnel will be available to speak with the patient's clinician at a local medical facility. Patients will return to WRAMC at 12 weeks for a follow-up evaluation of their symptoms, or they will be contacted by phone if unable to return to WRAMC for their 12 week evaluation. After the 12 week evaluation, patients will be tapered off sertraline or placebo over 2 weeks. Tapering and discontinuation of the study medication or placebo will be done on a gradual basis over the 2 weeks (e.g., If the patient is on 150 mg, s/he could take 100 mg for 1 week, 50 mg for one week, then D/C). If, following the 12 week evaluation, subjects have recurrent symptoms which are distressing to them, or believe they need medication to keep their symptoms from recurring, pharmacologic and nonpharmacologic treatments will be discussed with them. Patients will be offered appropriate treatment, including sertraline, if medically indicated. The blind will not yet be broken, that is, patients will not be able to learn if they were being treated with placebo or sertraline. Subjects will then be contacted by phone or seen at 3, 6, 9, and 12 months following their 12 week follow-up evaluation for an assessment of their symptoms and general level of functioning. If patients are in the area, these follow-up evaluation may be done in person.

   Concomitant medications:

   Patients with difficulty sleeping will be instructed in sleep hygiene, interviewed for possible deterrents to sleep induction, and encouraged to permit the test medication time to begin if depression is felt to contribute to the sleep disturbance. If difficulty initiating or maintaining sleep persist, Ambien 5-10 mg po qd (a non-serotoninergic hypnotic) will be offered. Benadryl 25-50 mg may also be considered for sleep induction. If clinically indicated, other medication may be prescribed.

   Patients with headaches will be counseled about precipitants in an attempt to maximize non-pharmacologic management of headache. If pain persists, enteric-coated ASA will be prescribed. For patients non-responsive to ASA (headache or other pain syndromes), non-steroidal antiinflammatory medications will be permitted. For vascular headaches, Midrin or sumatriptin may be used. If clinically indicated, other medication may be prescribed.

   If a patient has severe depression not responding to test article/placebo, and the treating physician deems antidepressant medication necessary, a non-SSRI medication, nortriptyline, will be used as the first line medication. Nortriptyline has been shown effective in post stroke depression (18), and may be monitored by plasma levels, thus being a good medication to combine with either placebo or sertraline. If nortriptyline is not effective (or if nortriptyline is not appropriate for that particular patient), the treating physician will chose whatever antidepressant is clinically indicated. Appropriate clinical care of the patient is the first priority.

   Pregnant women may not participate in this study. Women of childbearing age will take a urine or blood pregnancy test before starting this study to confirm they are not pregnant. As part of the informed consent, women are advised to avoid pregnancy for at least 6 weeks after receiving the drug treatment and will be advised about reliable methods of birth control. Breast-feeding women will also be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury patients within 6 months of injury.
* Traumatic brain injury with:

  * Minimum severity - TBI with post traumatic amnesia.
  * Maximum severity - recovery to a Rancho los Amigos (see Appendix II) level 7 or 8 by six months after injury.
* The C Criterion of DSM IV diagnosis of Post Concussive Disorder (PCD- Research Criteria), with symptoms persisting for a minimum of 4 weeks.
* Military beneficiary.

Exclusion Criteria:

* Severe prior neurologic or psychiatric illness, such as stroke or psychosis. (Previous nonpsychotic depression is not an exclusion criterion)
* Contraindication to the use of sertraline.
* Previous severe traumatic brain injury (defined as TBI with period of unconsciousness greater than 1 week prior. This exclusion refers only to TBI's prior to the current injury, which is within the past 6 months).
* Pregnancy
* Current active suicidal ideation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2000-02; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Gouvier-PCSC
Post Concussive Scale
Hamilton Depression Scale
Montgomery Asberg Depression Rating
Diagnosis of PCD by DSM-IV

SECONDARY OUTCOMES:
Smell Identification Test

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jaffee, MD, Study Director — The Defense and Veterans Brain Injury Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States